CLINICAL TRIAL: NCT05819528
Title: Primary Cardiac Lymphoma: Italian Multicenter Experience
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_Lympho-Heart
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Primary Cardiac Lymphoma
Keywords: PCL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — In order to perform pathology review, centers are requested to send all the histological and immunohistochemical slides performed at the local site for diagnosis and the block. A possible alternative to the block is 15 unstained slides. Only block and/or only unstained slides availability is not accepted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patients with a diagnosis primary cardiac lymphoma. The study includes patients with PCL diagnosed from 01/01/2000 to 31/12/2020.

SUMMARY:
The rationale of this study is to provide an overview on PCL (Primary Cardiac Lymphoma) in Italy, trying to shed light on unknown aspects of the disease and on unanswered questions about its management that could be helpful in clinical practice.

DETAILED DESCRIPTION:
Primary cardiac lymphoma (PCL), an extranodal lymphoma involving only the heart (with possible involvement of the pericardium) is a rare entity, accounting for 2% of primary cardiac tumors and 0.5% of extranodal lymphomas. It is more frequent in males; clinical presentation is predominated by cardiac symptoms. The most common histology is Diffuse Large B Cell Lymphoma (DLBCL). Being DLBCL the most frequent histology, patients are usually treated with R-CHOP (rituximab - cyclophosphamide, doxorubicin, vincristine and prednisone) or R-CHOP-like chemoimmunotherapy regimens, with an historically poor outcome, although in the last years survival rates significantly increased. Due to the rarity of this condition, isolated case reports and a few reviews have been published so far, that in most cases included a population collected in a wide period of time, heterogeneously managed both in terms of treatments received and follow-up, and who often did not strictly respect the criteria of PCL. Indeed, while some aspects of PCL are well-known, especially the ones concerning its clinical presentation, a few topics deserve more in-depth analysis. The rationale of this study is to provide an overview on PCL in Italy, trying to shed light on unknown aspects of the disease and on unanswered questions about its management that could be helpful in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCL (any histotype) defined as an extranodal lymphoma involving only the heart with possible involvement of the pericardium.
* Age ≥18 years.
* Diagnosis histologically confirmed. Cytofluorimetry analysis of pericardial fluid showing phenotypic features consistent with a primary cardiac lymphoma is permitted if a biopsy sample is not feasible/available for diagnosis; monoclonality is not accepted as a surrogate for diagnosis.
* Date of diagnosis: from 1st January 2000 to 31st December 2020.
* Only patients treated in first-line with chemoimmunotherapy regimens including an anti-CD20 monoclonal antibody are eligible for the study.
* Signed written informed consent (in case of unreachable subject please see chapter 11.2)

Exclusion Criteria:

* Secondary cardiac involvement from lymphoma; primary mediastinal lymphoma with pericardial infiltration or other lymphomas with involvement of the pericardium/the heart by contiguity and primary effusion lymphoma are not included in this study.
* Patients treated with chemotherapy regimens that did not include an anti-CD20 monoclonal antibody as first-line therapy.
* Refuse to sign a written informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient affected by primary cardiac lymphoma from 1st January 2000 to 31st December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | The endpoint will be evaluated within 2 months from the end of data collection. The end of data collection is scheduled within the Q4 (fourth quarter) of 2023.
  Overall survival, the percentage of patients alive of the cohort (patients with cardiac lymphoma diagnosed from 01/01/2000 to 31/12/2020).

SECONDARY OUTCOMES:
Complete remission (CR) | The endpoint will be evaluated within 2 months from the end of data collection. The end of data collection is scheduled within the Q4 (fourth quarter) of 2023.
  The Complete Remission is defined as the lack of detectable evidence of tumor in the cohort of patients (patients with cardiac lymphoma diagnosed from 01/01/2000 to 31/12/2020).
Overall Response Rate (ORR) | The endpoint will be evaluated within 2 months from the end of data collection. The end of data collection is scheduled within the Q4 (fourth quarter) of 2023.
  The Overall Response Rate is defined as the proportion of patients who have a partial or complete response to therapy (patients with cardiac lymphoma diagnosed from 01/01/2000 to 31/12/2020).
Progression-Fee Survival (PFS) | The endpoint will be evaluated within 2 months from the end of data collection. The end of data collection is scheduled within the Q4 (fourth quarter) of 2023.
  The Progression-Free Survival is the length of time during and after the treatment that patients live with the disease, but it does not get worse (patients with cardiac lymphoma diagnosed from 01/01/2000 to 31/12/2020).
Frequencies of the type of chemo(immuno)therapy and of the number of cycles received as first and second line. | The endpoint will be evaluated within 2 months from the end of data collection. The end of data collection is scheduled within the Q4 (fourth quarter) of 2023.
  The numbers of treatment types and numbers of cycles of therapy received by the cohort of patients (patients with cardiac lymphoma diagnosed from 01/01/2000 to 31/12/2020).
Frequencies of the type of Central Nervous System (CNS) prophylaxis | The endpoint will be evaluated within 2 months from the end of data collection. The end of data collection is scheduled within the Q4 (fourth quarter) of 2023.
  The numbers of treatment prophylaxis types for Central Nervous System administered to the cohort of patients (patients with cardiac lymphoma diagnosed from 01/01/2000 to 31/12/2020).
Cumulative incidence rate of Central Nervous System (CNS) relapse detected during treatment or follow-up. | The endpoint will be evaluated within 2 months from the end of data collection. The end of data collection is scheduled within the Q4 (fourth quarter) of 2023.
  The proportion of patients with disease relapse on Central Nervous System (CNS)
Characteristics of patients | The endpoint will be evaluated within 2 months from the end of data collection. The end of data collection is scheduled within the Q4 (fourth quarter) of 2023.
  Analysis of the following characteristics: Age, gender, disease localization (atria, ventricles, cardiac arteries and veins, pericardium), HIV positivity, type of symptoms at diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Lucchini, MD, Principal Investigator — Trieste - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia
Locations (17):
- Italy (17):
  - Presidio ospedaliero "A. TORTORA" - U.O. Onco-ematologia, Pagani, Salerno
  - AOU di Sassari - Ematologia, Sassari, SS
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia, Trieste, TS
  - Ospedale Dell'angelo - U.O. Ematologia, Mestre, Venezia
  - Azienda Ospedaliera Papa Giovanni XXIII - Ematologia, Bergamo
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna - Ematologia e fisiopatologia della coagulazione, Ferrara
  - Istituto Scientifico San Raffaele - Unitа Linfomi - Dipartimento Oncoematologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano - Ematologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - Ospedale S. Maria della Misericordia - Ematologia, Perugia
  - AOU Pisana - U.O. Ematologia, Pisa
  - Roma - Universitа Cattolica S. Cuore - Ematologia, Roma
  - AO Sant'Andrea - Ematologia, Roma
  - A.O. S. Maria di Terni - S.C. Oncoematologia, Terni
  - A.O.U. Città della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - AOU Integrata di Verona - U.O. Ematologia, Verona

IPD SHARING:
Plan to Share IPD: No